CLINICAL TRIAL: NCT03934502
Title: Phase I, Open-Label, Randomized, Single-Dose, Four-Period, Four-Sequence Crossover Study to Compare the Effects of a Light Meal and of a Low-Fat Meal Timing on Evobrutinib Bioavailability in Healthy Volunteers
Brief Title: Effect of Meal Composition and Timing on Evobrutinib Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200527_0072; 2019-000877-21 (EudraCT Number); NCT04200430 (obsolete NCT alias)
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Evobrutinib; Pharmacokinetics
MeSH Terms: interventions — evobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Evobrutinib: Treatment Sequence A, B, C, D (Experimental): Participant will receive single oral dose of evobrutinib after an overnight fast of at least 10 hours (Treatment A) for 3 days, followed by within 30 minutes after start of a light meal (Treatment B) for 2 days, followed by 1 hour prior to a low-fat meal (Treatment C) for 2 days, followed by 2 hours after start of low-fat meal (Treatment D) for 2 days. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Treatment Sequence B, D, A, C (Experimental): Participant will receive single oral dose of evobrutinib within 30 minutes after start of a light meal (Treatment B) for 3 days, followed by 2 hours after start of a low-fat meal (Treatment D) for 2 days, followed by after an oversight fast of at least 10 hours (Treatment A) for 2 days, followed by 1 hour prior to a low-fat meal (Treatment C) for 2 days. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Treatment Sequence C, A, D, B (Experimental): Participant will receive single oral dose of evobrutinib 1 hour prior to a low-fat meal (Treatment C) for 3 days, followed by after an oversight fast of at least 10 hours (Treatment A) for 2 days, followed by 2 hours after start of a low-fat meal (Treatment D) for 2 days followed by within 30 minutes after start of a light meal (Treatment B) for 2 days. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Treatment Sequence D, C, B, A (Experimental): Participant will receive single oral dose of evobrutinib 2 hours after start of a low-fat meal (Treatment D) for 3 days, followed by 1 hour prior to a low-fat meal (Treatment C) for 2 days, followed by within 30 minutes after start of a light meal (Treatment B) for 2 days, followed by after an overnight fast of at least 10 hours (Treatment A) for 2 days. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Evobrutinib

INTERVENTIONS:
Drug: Evobrutinib — Participants will receive single oral dose of evobrutinib either after an overnight fast of at least 10 hours (Treatment A), within 30 minutes after start of a light meal (Treatment B), 1 hour prior to a low-fat meal (Treatment C), or 2 hours after start of a low-fat meal (Treatment D).
  Other Names: M2951

SUMMARY:
This study will evaluate the Pharmacokinetics (PK) of the Phase II tablet formulation of Evobrutinib under fasted conditions, within 30 minutes after start of a light meal, one hour prior to start of a low-fat meal, and 2 hours after start of a low-fat meal.

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy as medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring
* Participants are stable non-smokers for at least 3 months preceding screening
* Male or female participants agree to be consistent with local regulations on contraception methods
* Female participants are not pregnant or breastfeeding, and at least one of the following condition applies:
* Not a woman of childbearing potential (WOCBP) or
* If a WOCBP, use a highly effective contraceptive method (that is, with a failure rate of less than (<) 1 percent per year, preferably with low user dependency for the following time period:
* Before the first dose of the study intervention, if using hormonal contraception:
* Has completed at least one 4-week cycle of an oral contraception pill and either had or has begun her menses or
* Has used a depot contraceptive or extended-cycle oral contraceptive for least 28 days and has a documented negative pregnancy test using a highly sensitive assay and
* A barrier method
* During the intervention period
* After the study intervention period (that is after the last dose of study intervention is administered) for at least 90 days, plus 30 days (a menstrual cycle) after the last dose of study intervention and agree not to donate eggs (ova, oocytes) for reproduction during this period. The Investigator evaluates the effectiveness of the contraceptive method in relationship to the first dose of study intervention
* Females have a negative serum pregnancy test at the Screening Visit and within 24 hours before the first dose of study intervention If a urine test cannot be confirmed as negative (example: an ambiguous result), a serum pregnancy test is required
* The Investigator reviews the medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a female with an early undetected pregnancy
* Male participants should agree to the following during the study intervention period and for at least 3 months
* after the last dose of study intervention:
* Refrain from donating sperm,
* plus either:
* Abstain from intercourse with a female, Or
* use a male condom:
* When having sexual intercourse with a WOCBP, who is not currently pregnant, and advise her to use a highly effective contraceptive method with a failure rate of <1 percent per year, since a condom may break or leak
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Prior history of cholecystectomy or splenectomy, and any clinically relevant surgery within 6 months prior to screening
* History of any malignancy
* History of chronic or recurrent acute infection or any bacterial, viral, parasitic or fungal infections within 30 days prior to screening and at any time between screening and admission, or hospitalization due to infection within 6 months prior to screening
* History of shingles within 12 months prior to screening
* History of drug hypersensitivity, ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients
* History of alcoholism or drug abuse within 2 years prior to screening, or evidence of such abuse as indicated by the laboratory assays conducted during screening
* History of residential exposure to tuberculosis, or a positive QuantiFERON® test within 4 weeks prior to screening
* Administration of live vaccines or live-attenuated virus vaccines within 3 months prior to screening
* Any condition, including findings in the laboratory tests, medical history, or other screening assessments, that in the opinion of the Investigator constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study's objectives, conduct, or evaluation
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Evobrutinib | Pre-dose up to 24 hours post-dose
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUC0-inf) of Evobrutinib | Pre-dose up to 24 hours post-dose
Maximum Plasma Concentration Observed (Cmax) of Evobrutinib | Pre-dose up to 24 hours post-dose

SECONDARY OUTCOMES:
Number of Participants With Treatment -Emergent Adverse Events (TEAEs) | Day 1 up to Day 9
Number of Participants With Clinically Significant Change From Baseline in Vital Signs, Laboratory Parameters and Electrocardiogram Findings | Day 1 up to Day 9
  Number of participants with clinically significant change from baseline in vital signs, laboratory parameters and electrocardiogram findings will be reported
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 24 Hours After Drug Administration (AUC0-24) of Evobrutinib | Pre-dose up to 24 hours post-dose
Area Under The Concentration-Time Curve from Time Zero to Time 12 Hours (AUC0-12) of Evobrutinib | Pre-dose up to 12 Hours post-dose
Time to Reach Maximum Concentration (Tmax) of Evobrutinib in Plasma | Pre-dose up to 24 hours post-dose
Time Prior to the First Measurable (non-zero) Concentration of Evobrutinib | Pre-dose up to 24 hours post-dose
Apparent Elimination Half Life (t1/2) of Evobrutinib | Pre-dose up to 24 hours post-dose
Apparent Clearance (CL/f) of Evobrutinib | Pre-dose up to 24 hours post-dose
Apparent Volume of Distribution During Terminal Phase (VZ/f) of Evobrutinib | Pre-dose up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt Germany, an affiliate of Merck KGaA, Darmstadt, Germany will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0072
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html